CLINICAL TRIAL: NCT04666909
Title: Take the Pressure Off, NYC! Staten Island Barbershop Initiative
Brief Title: Take the Pressure Off, NYC!
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-00978
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertension Group: Participants will receive a free blood pressure screening and receive educational counseling about the importance of maintaining a healthy blood pressure. In addition, educational counseling will be administered in months 3 and 6.
  Interventions: Diagnostic Test: blood pressure

INTERVENTIONS:
Diagnostic Test: blood pressure — The Welch Allyn ABPM 7100 is an easy-to-use 24-hour ambulatory blood pressure monitor that is designed to help avoid the effects of white coat hypertension, provide accurate sleep blood pressure readings, and tailor drug therapy regimes to your individual patient's needs.
  This device is programmed to take three BP readings a minute apart. To be eligible, participants must have an average SBP > 135 mm Hg or DBP > 85 mmHg (based on the average of 3 BP readings); or average SBP > 130 mm Hg or DBP > 80 mm hg (for those with diabetes or kidney disease) based on JNC-7 criteria for uncontrolled HTN.
  Other Names: ABPM 7100 Ambulatory Blood Pressure Monitor

SUMMARY:
Briefly, a trained barbershop navigator will work with each barbershop to measure blood pressure on each adult customer who agrees, and to provide culturally-targeted education about high blood pressure and its consequences, and motivational interviewing-informed counseling about therapeutic lifestyle changes. For customers found to have high blood pressure, the navigator will also provide referral and navigation to a medical provider and, as appropriate, a local pharmacy.

DETAILED DESCRIPTION:
This program will be patterned after barbershop-based blood pressure programs that have demonstrated efficacy in achieving lower blood pressure and improved hypertension control rates among Black men with high blood pressure. This program will reach 10-12 barbershops per year, working with 2-3 barbershops each quarter. Briefly, a trained barbershop navigator will work with each barbershop t o measure blood pressure on each adult customer who agrees, and to provide culturally-targeted education about high blood pressure and its consequences, and motivational interviewing-informed counseling about therapeutic lifestyle changes. For customers found to have high blood pressure, the navigator will also provide referral and navigation to a medical provider and, as appropriate, a local pharmacy. At all recruitment events, all study team members and potential participants must wear masks and practice social distancing when appropriate. Participants who do not have face masks should be offered masks for continued outreach participation. Study team members will also wear gloves and have hand sanitizer visible. When available, staff should wash hands frequently with soap and water. If this option is not available, staff should frequently use hand sanitizer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age 18 years or older
* Self-identified as a black or African American male
* Have uncontrolled hypertension defined as SBP>135 mmHg or DBP>85 mmHg and SBP >130 mmHg or DBP >80 mmHg (in those with diabetes) at the screening

Exclusion Criteria:

* Under the age of 18
* Does not consent to participate

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Black men will be recruited for this study which is a group that is often underrepresented in cardiovascular (CVD) risk reduction and in clinical practices
Study Population: This study is limited to men. Because the goal of this study is to reduce the racial disparities in hypertension-related outcomes between minority ethnic/racial groups and whites, the participants in this study will be self-identified as African American or Black
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure over 6 months | Initial Study Day 1, Follow up 1 (Day 90 +/- 10), Follow up 2 ((Day 180+/-10)
  Blood pressure will be measured with FDA approved blood pressure monitor on the first day of the study, 3 months and 6 months after the initial study day.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ravenell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: This data will not be available outside of the study team and our partners
Access Criteria: The investigator who proposed to use the data.